CLINICAL TRIAL: NCT03237338
Title: The Study of Brain GABA and Brain Functional Modulatory Mechanism of Chronic Insomnia Disorder Using Acupuncture at "Combined Magical-door" Acupoints
Brief Title: The Study of Mechanism of Chronic Insomnia Disorder Using Acupuncture Based on Changes of Brain GABA and fMRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongfang Hospital Beijing University of Chinese Medicine (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2017-JYB-JS-166
Record Dates: First submitted 2017-07-24; First posted 2017-08-02 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2020-08

CONDITIONS: Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insomnia-ture acupuncture (Experimental): True acupuncture at the "Magical-door", "Si-shen-cong", "Shen-ting", "Local-cave" acupoints will be administered on CID patients Intervention: Procedure: true acupuncture
  Interventions: Procedure: ture acupuncture
- Insomnia-sham acupuncture (Sham Comparator): Sham acupuncture at the "Magical-door", "Si-shen-cong", "Shen-ting", "Local-cave" acupoints will be administered on CID patients Intervention: Procedure: true acupuncture
  Interventions: Procedure: sham acupuncture

INTERVENTIONS:
Procedure: ture acupuncture — ture acupuncture at the "Magical-door", "Si-shen-cong", "Shen-ting", "Local-cave" acupoints, three times per week and last for 6 weeks
  Arms: Insomnia-ture acupuncture
Procedure: sham acupuncture — Sham acupuncture at the "Magical-door", "Si-shen-cong", "Shen-ting", "Local-cave" acupoints, three times per week and last for 6 weeks
  Arms: Insomnia-sham acupuncture

SUMMARY:
Insomnia disorder is one of the major neuropsychiatric diseases which received more attention in recent years. Disturbances in the amino acid neurotransmitter, gama-amino butyric acid (GABA) and hyperarousal of cortex are hypothesized to contribute to the neurobiology of insomnia. Both animal experiment and clinical observation have demonstrated that acupuncture can generate treatment effect on insomnia symptom. However, the underlying mechanism remains unclear. The principal objective of this project is to use magnetic resonance spectroscopy (MRS) as well as acupuncture to provide the first in vivo characterization of cortical GABA levels between pro- and post-acupuncture treatment in individuals with chronic insomnia disorder (CID), and use resting state functional magnetic resonance imaging (fMRI) to determine whether CID patients have altered brain connectivity and network parameter changes. The investigators are also exploring the correlation between cortical GABA levels, fMRI parameter changes and abnormalities in sleep parameters and neuropsychology test in CID patients.

DETAILED DESCRIPTION:
Three groups of subjects (CID accepted true acupuncture, CID accepted sham acupuncture and healthy) will participate in the study. All subjects will undergo a laboratory blood test, physical and neurological examination, polysomnography (PSG) and an extensive battery of neuropsychological assessments. All subjects meeting eligibility criteria for the study will complete a baseline MRS and fMRI to evaluate differences in multi-modality brain GABA and fMRI parameters between the patients and healthy. After randomized acupuncture treatment, investigators will compare brain metabolic and functional parameters to elucidate the neural mechanism of acupuncture therapy on insomnia, provide theoretical evidence from the perspective of neurotransmitters and brain network.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic insomnia disorder (CID) met the criteria of the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
* Subject has history of chronic insomnia (difficulty with sleep induction, awakenings during the night, early morning awakening) of at least 3 months
* Must be able to cooperate with cognitive testing and MRI scan

Exclusion Criteria:

* Known pre-existing sleep disorder other than chronic insomnia disorder
* Circadian rhythm sleep disorder determined by sleep-wake cycles of sleep (such as work time at day and night alternation)
* Severe general medical disorders of cardiovascular, endocrine, renal, or hepatic systems
* Clinical diagnosis of AD or Parkinson's neurodegenerative diseases
* Moderate or severe psychological illness
* Clinical history of stroke or other severe cerebrovascular disease
* Clinical history of malignancies disease
* Active treatment with antipsychotic medications, benzodiazepines or other hypnotic agents (i.e. Trazodone, Mirtazapine, Zolpidem, Zaleplon)
* Alcohol or drug abuse

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-12-26 (Actual); Primary Completion 2021-08-20 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
change from baseline brain GABA level at 24 days | at the 2 day before acupuncture treatment and the 24th day after acupuncture treatment
  GABA levels in the prefrontal gyrus, occipital gyrus

SECONDARY OUTCOMES:
brain functional connectivity | at the 24th day after acupuncture treatment
  functional connectivity between the medial prefrontal cortex and other brain regions
Wake time after sleep onset (WASO) | at the 24th day after acupuncture treatment
  WASO is the total time of awake occurring between sleep onset and final wake up

CONTACTS AND LOCATIONS:
Locations (1):
- Dongfang Hospital Affiliated to Beijing University of Chinese Medicine, Beijing, China